CLINICAL TRIAL: NCT02834039
Title: Comparison of Ventilation Distribution Between Tidal Volume 6ml/kgBW and 10ml/kgBW in Laparoscopic Nephrectomy Patients
Brief Title: Comparison of Ventilation Distribution Between Tidal Volume 6ml/kgBW and 10ml/kgBW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, Consultant, Anesthesiologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes004
Record Dates: First submitted 2016-07-12; First posted 2016-07-15 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Laparoscopic Nephrectomy
Keywords: Tidal volume; renal transplant; donor; nephrectomy; ventilation; Living renal transplant donor patient
MeSH Terms: conditions — Respiratory Aspiration | interventions — Tidal Volume

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Tidal volume 6 ml/kgBW (Active Comparator): Tidal volume 6 ml/kgBW was given to patients after endotracheal tube was inserted properly
  Interventions: Procedure: Tidal volume 6 ml/kgBW
- Tidal volume 10 ml/kgBW (Active Comparator): Tidal volume 10 ml/kgBW was given to patients after endotracheal tube was inserted properly.
  Interventions: Procedure: Tidal volume 10 ml/kgBW

INTERVENTIONS:
Procedure: Tidal volume 6 ml/kgBW — Tidal volume 6ml/kgBW was given to subjects after endotracheal tube was inserted properly.
  Arms: Tidal volume 6 ml/kgBW
Procedure: Tidal volume 10 ml/kgBW — Tidal volume 10 ml/kgBW was given to subjects after endotracheal tube was inserted properly.
  Arms: Tidal volume 10 ml/kgBW

SUMMARY:
This study aims to compare the ventilation Distribution between tidal Volume 6ml/kgBW and tidal volume 10ml/kgBW in laparoscopic nephrectomy patients

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine University of Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study. Non-invasive blood pressure (NIBP) monitor, electrocardiogram (ECG) and pulse-oximeter was set on the subjects in the operation room. Anesthesia procedure was epidural regional block. After given premedication (midazolam 0.05 mg/kgBW and fentanyl 1-2 ug/kgBW), induced with propofol, 1-2 mg/kgbb, endotracheal tube intubation was done facilitated by atracurium 0.5 mg/kgbb. Mechanical ventilation was set up with volume control mode, (Positive End Expiratory Pressure) PEEP 5cmH2O (5 centimeters of water), O2 fraction (FiO2) 30-50%, target carbondioxide (CO2) 35-45%. Volume tidal was given according to the group (6 mL/kgBW or 10 ml/kgBW). Hemodynamic, ventilation parameter, Electrical Impedance Tomography (EIT) parameter were recorded. If desaturation happened intraoperatively will be managed by increasing FiO2 and recruitment maneuver until oxygen saturation (SpO2) >95%. Data was analyzed using Statistical Program for Social Sciences (SPSS), for numeric data using unpaired T-test or Mann-Whitney-U test, for categorical data using Chi-square or Fisher Exact Test. Significant value is p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-60 years old
* Subjects with good health condition (did not suffer from cancer, diabetes mellitus, kidney diseases, cardiovascular diseases, liver diseases, hematologic disorders, HIV, hepatitis)
* Subjects had the same blood type with the renal recipients and had passed cross match test
* Subjects were willing to be renal donors.

Exclusion Criteria:

* Subjects with pulmonary diseases or PaO2 (arterial partial pressure of oxygen) /FiO2 < 300 mmHg
* Subjects with Body Mass Index (BMI) > 30 kg/m2
* Subjects who had mechanical ventilation 2 weeks prior to the surgery
* Subjects with congestive heart failure
* Subjects with neuromuscular diseases.

Drop out criteria:

* Subjects with intraoperative pulmonary complications not due to ventilation
* Subjects with intraoperative cardiac arrest
* Subjects with desaturation that could not be managed by FiO2 increase, PEEP or recruitment maneuver, and required tidal volume changes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2017-02-28 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Tidal impedance variation regional (TIV-ROI) | 2 months
  Evaluating ROI values displayed on EIT Dräger PulmoVista® 500 monitor.
Global End expiratory lung impedance difference (ΔEELI-g) | 2 months
  Global End expiratory lung impedance difference (ΔEELI-g) will be measured by the EIT monitor.
Regional End expiratory lung impedance difference (ΔEELI- ROI) | 2 months
  Regional End expiratory lung impedance difference (ΔEELI-g) will be measured by the EIT monitor.
Compliance regional (CR) | 2 months
  Tidal Impedance Variation value divided by atmospheric pressure above PEEP value.

CONTACTS AND LOCATIONS:
Overall Officials: Dita Aditianingsih, Consultant, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jha V, Garcia-Garcia G, Iseki K, Li Z, Naicker S, Plattner B, Saran R, Wang AY, Yang CW. Chronic kidney disease: global dimension and perspectives. Lancet. 2013 Jul 20;382(9888):260-72. doi: 10.1016/S0140-6736(13)60687-X. Epub 2013 May 31. PMID 23727169
- [Background] Rizzotti L, Vassiliou M, Amygdalou A, Psarakis Ch, Rasmussen TR, Laopodis V, Behrakis P. Respiratory system mechanics during laparoscopic cholecystectomy. Respir Med. 2002 Apr;96(4):268-74. doi: 10.1053/rmed.2001.1264. PMID 12000007
- [Background] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482
- [Background] Ricard JD, Dreyfuss D, Saumon G. Ventilator-induced lung injury. Eur Respir J Suppl. 2003 Aug;42:2s-9s. doi: 10.1183/09031936.03.00420103. PMID 12945994
- [Background] de Prost N, Ricard JD, Saumon G, Dreyfuss D. Ventilator-induced lung injury: historical perspectives and clinical implications. Ann Intensive Care. 2011 Jul 23;1(1):28. doi: 10.1186/2110-5820-1-28. PMID 21906379
- [Background] Costa EL, Lima RG, Amato MB. Electrical impedance tomography. Curr Opin Crit Care. 2009 Feb;15(1):18-24. doi: 10.1097/mcc.0b013e3283220e8c. PMID 19186406
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Moerer O, Hahn G, Quintel M. Lung impedance measurements to monitor alveolar ventilation. Curr Opin Crit Care. 2011 Jun;17(3):260-7. doi: 10.1097/MCC.0b013e3283463c9c. PMID 21478747
- [Background] Victorino JA, Borges JB, Okamoto VN, Matos GF, Tucci MR, Caramez MP, Tanaka H, Sipmann FS, Santos DC, Barbas CS, Carvalho CR, Amato MB. Imbalances in regional lung ventilation: a validation study on electrical impedance tomography. Am J Respir Crit Care Med. 2004 Apr 1;169(7):791-800. doi: 10.1164/rccm.200301-133OC. Epub 2003 Dec 23. PMID 14693669
- [Background] Riera J, Riu PJ, Casan P, Masclans JR. [Electrical impedance tomography in acute lung injury]. Med Intensiva. 2011 Nov;35(8):509-17. doi: 10.1016/j.medin.2011.05.005. Epub 2011 Jun 15. Spanish. PMID 21680060
- [Background] Lorenzo AJ, Karsli C, Halachmi S, Dolci M, Luginbuehl I, Bissonnette B, Farhat WA. Hemodynamic and respiratory effects of pediatric urological retroperitoneal laparoscopic surgery: a prospective study. J Urol. 2006 Apr;175(4):1461-5. doi: 10.1016/S0022-5347(05)00668-3. PMID 16516022
- [Background] Goncalves LO, Cicarelli DD. Alveolar recruitment maneuver in anesthetic practice: how, when and why it may be useful. Rev Bras Anestesiol. 2005 Dec;55(6):631-8. doi: 10.1590/s0034-70942005000600006. English, Portuguese. PMID 19468537